CLINICAL TRIAL: NCT04820283
Title: Early Interventions for Primary Care Patients With Stress-related Ill-health: a Randomized Controlled Non-inferiority Trial of a Collaborative Care Intervention vs. Cognitive Behavior Therapy
Brief Title: Early Interventions for Primary Care Patients With Stress-related Ill-health: a Non-inferiority RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Erik Hedman, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Early interventions for stress
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stress
MeSH Terms: interventions — Nurses

STUDY DESIGN:
Intervention Model Description: Randomized controlled non-inferiority trial with two arms. A non-inferiority margin of Cohen's d 0.3 on the primary outcome Perceived Stress Scale at post-treatment (change from baseline to 12 weeks) will be used. For test of non-inferiority on the primary outcome, a one-sided 95% confidence interval (CI) will be used. If the two-sided 95% CI (exploratory analyses) does not include 0 this will be interpreted as indicating superiority of the corresponding treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Care manager intervention (nurse) (Experimental)
  Interventions: Behavioral: Care manager intervention (nurse)
- Internet-based CBT (Active Comparator)
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: Care manager intervention (nurse) — In this intervention, a primary care nurse provides the participant with self-management support to manage stress-related problems. The participant meets with the nurse face-to-face for typically 2 to 6 sessions.
  Arms: Care manager intervention (nurse)
Behavioral: CBT — In this intervention, the participant receives therapist supported self-help CBT. The participant randomized to this arm can choose to receive the treatment via an online treatment platform or via bibliotherapy, i.e., a self-help book.The treatment is comprised of 12 modules or chapters, which entail information about stress management techniques including behavioral activation and exposure. The participant that chooses online CBT is guided by a therapist who provides feedback on homework assignments through written asynchronous text messages; the patient who chooses bibliotherapy is guided by a therapist in typically 2 to 5 face-to-face sessions at a primary care clinic.
  Arms: Internet-based CBT

SUMMARY:
Stress-related ill-health is rated one of the largest health challenges in the western world. The most empirically supported treatment for stress-related disorders is cognitive behaviour therapy (CBT), but accessibility is low and most patients in primary care do not receive this evidence-based treatment. Collaborative care has been shown to be an effective working model for primary care patients with mental health problems. This type of care intervention has however not been compared against CBT, which is arguably the gold standard treatment for this patient group. The overarching purpose of this project is to investigate if implementation of two treatment models - collaborative care and therapist-guided self-help CBT -can be effective as early interventions for primary care patients with stress-related ill-health.

DETAILED DESCRIPTION:
Stress-related ill-health is rated one of the largest health challenges in the western world. The most empirically supported treatment for stress-related disorders is cognitive behaviour therapy (CBT), but accessibility is low and most patients in primary care do not receive this evidence-based treatment. Collaborative care has been shown to be an effective working model for primary care patients with mental health problems. In this study collaborative care is conducted by a nurse who provides the patient with self-management support. This intervention has been implemented at Gustavsbergs primary care clinic in Stockholm as a means to increase accessibility and quality of care for the large group of patients with stress-related ill-health. This type of care intervention has however not been compared against CBT, which is arguably the gold standard treatment for this patient group.

Our research group has developed and tested a therapist-guided self-help CBT (SH-CBT) that can be delivered online or as a self-help book with support by a clinician for stress-related ill health, which has been shown to be effective and also potentially very suitable for the primary care context. The overarching purpose of this project is to investigate if implementation of two treatment models - collaborative care and SH-CBT - can be effective as early interventions for primary care patients with stress-related ill-health.

Main research question: Is a brief collaborative care intervention provided by a nurse at least as effective as SH-CBT delivered by a psychologist for primary care patients with mild to moderate symptoms of stress?

Note: In may 2022, the research group made revisions to the study procedures in terms of administration format of CBT and inclusion criteria. These specific changes were made: (1) Participants randomized to SH-CBT are allowed to choose if they want to receive the treatment as therapist-guided online CBT or as therapist-guided bibliotherapy CBT. Participants are exposed to the same treatment content, but in the former case the material is presented on a secure website with asynchronous written therapist support and in the latter case the content is provided through a self-help book and the participant has 2-5 face-to-face appointments with the therapist; (2) It is no longer required that participants has adjustment disorder, instead participants have to have (a) a score on the Perceived Stress Scale-10 of 20 or higher, (b) stress-related ill-health as their principal problem, and (c) a duration of their problems of at least 1 month; (3) The sick-leave criterion is changed so that participants to be included are allowed to have been on full time sick-leave for maximum 2 months (instead of 50% for maximum 1 month).

The revisions described above were made in order to better operationalize the patient population "patients with mild to moderate stress-related ill-health" and to increase the recruitment of participants to the study. When the revisions were implemented approximately 20 participants had been included in the study. The revisions were approved by the Swedish Ethical Review Authority (ID 2022-00990-02).

Note 2: In the autumn of 2023, a new power calculation was conducted where full use of the 5 assessment points between baseline and post-treatment (12 weeks) was taken into account. This new power calculation, based in linear mixed models analysis for longitudinal data, showed that in order to have 80% power to demonstrate non-inferiority (non-inferiority margin d=0.3; one-sided 95% confidence interval) given a true effect difference of 0, approximately 170 participants (85 per treatment arm) will be needed.

ELIGIBILITY:
Inclusion Criteria:

* At least 16 years of age
* A score of 20 or higher on the Perceived Stress Scale-10
* Stress-related ill-health is the principal problem
* Duration of problems for at least 1 month
* Have symptoms in the mild to moderate range
* Be able to read and write in Swedish
* Have access to a computer with Internet connection
* If the participant is on sick leave then the sick leave period should have a maximum duration of 2 months (full time sick-leave for 2 months is thus allowed)

Exclusion Criteria:

* Ongoing other psychological treatment for stress-related problems

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | Baseline, weeks 3, 6, 9, 12 (post-treatment), 1-year follow-up
  Change in PSS at post-treatment and follow-up compared to baseline (scale range 0-40, higher score means more symptoms)

SECONDARY OUTCOMES:
Shirom-Melamed Burnout Questionnaire (SMBQ) | Baseline, weeks 3, 6, 9, 12 (post-treatment), 1-year follow-up
  Change in SMBQ at post-treatment and follow-up compared to baseline (scale range 1-7, higher score means more symptoms)
Insomnia Severity Index (ISI) | Baseline, weeks 3, 6, 9, 12 (post-treatment), 1-year follow-up
  Change in ISI at post-treatment and follow-up compared to baseline (scale range 0-28, higher score means more symptoms)
Generalized Anxiety Disorder-7 (GAD-7) | Baseline, week 12 (post-treatment), 1-year follow-up
  Change in GAD-7 at post-treatment and follow-up compared to baseline (scale range 0-21, higher score means more symptoms)
Patient Health Questionnaire-9 (PHQ-9) | Baseline, weeks 3, 6, 9, 12 (post-treatment), 1-year follow-up
  Change in PHQ-9 at post-treatment and follow-up compared to baseline (scale range 0-27, higher score means more symptoms)
Brunnsviken Brief Quality of Life Index (BBQ) | Baseline, week 12 (post-treatment), 1-year follow-up
  Change in BBQ at post-treatment and follow-up compared to baseline (scale range 0-96, higher score means higher quality of life)
EuroQol 5D (EQ5D) | Baseline, week 12 (post-treatment), 1-year follow-up
  Change in EQ5D at post-treatment and follow-up compared to baseline (the answers will be converted to utility score of health states ranging from 0 to 1 where 0 represents death and 1 full health)
Trimbos and Institute of Medical Technology Assessment of Cost Questionnaire for Psychiatry (TIC-P) | Baseline, week 12 (post-treatment), 1-year follow-up
  The TIC-P enables estimation of costs by collecting information about participant resource utilization and costs related to production loss. Change in costs will be analyzed at post-treatment and follow-up compared to baseline.
Sick leave | 1 year from baseline
  Sick leave data from the Microdata for Analysis of Social Security (MiDAS) registry. Analyzed as full day equivalents.

OTHER OUTCOMES:
Credibility Scale (C-Scale) | Week 3
  Week 3 point estimate of treatment credibility rating (scale range 0-50, higher score means higher credibility)
Client Satisfaction Questionnaire-8 (CSQ-8) | week 12 (Post-treatment)
  Post-treatment point estimate of satisfaction with treatment (scale range 8-32, higher score means higher satisfaction with treatment)
Recovery Experience Questionnaire Short (REQ-S): putative mediator | Baseline, weeks 3, 6, 9, 12 (post-treatment)
  Change in REQ-S at post-treatment compared to baseline (scale range 0-28, higher score means more recovery)
Negative Events Questionnaire (NEQ-20) | Week 12 (post-treatment)
  Post-treatment estimate of potential negative events during treatment (scale range 0-80 where higher score means more negative events)
Adjustment Disorder New Module-8 (ADNM-8) | Baseline
  Point estimate at baseline for screening purposes (scale range 8-32 where higher score means more symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Gustavsbergs Primary Care Center, Gustavsberg, Stockholm County, Sweden